CLINICAL TRIAL: NCT03765684
Title: Effects of Various Parental and Gestational Factors on Offspring Body Composition and Health in Later Life in Helsinki Birth Cohort 2018-2022
Brief Title: Factors Affecting Newborn Body Composition and Later Health in Helsinki Birth Cohort 2018-2022
Acronym: HeBiCo
Status: Active, not recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Finnish Institute for Health and Welfare (Other Government); UKK Institute (Other)
Responsible Party: Principal Investigator, Saila Koivusalo, Associate Professor, Development Manager, Helsinki University Central Hospital
Other Study IDs: HUS/180/2018, HUS/512/2019
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Offspring, Adult; Lifestyle; Obesity, Childhood; Pregnancy Related; Child Development
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal and umbilical cord blood sample is collected and stored for later analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In Helsinki Birth Cohort 2018-2022 a large, longitudinal and well-phenotyped birth cohort of infants and their parents will be established. Mothers, fathers/spouses and their children in Helsinki and Uusimaa Hospital District are recruited in the study and newborn composition of the children born in Helsinki Women's Hospital will be measured. Data on maternal and paternal diet quality, physical activity and depression during and after pregnancy will be collected and data from the hospital and national registers will be collected. Health of offspring and parents will be followed during their later life.

DETAILED DESCRIPTION:
Helsinki Birth Cohort 2018-2022 (HeBiCo) study is designed to find evidence between various intrauterine exposures and offspring adiposity and later health. It will be examined how different maternal (e.g. chronic diseases, ethnicity, BMI), and obstetric factors (e.g. gestational weight gain, diagnoses during pregnancy) as well as parental lifestyle and psychological aspects (e.g. diet quality, physical activity, depression and anxiety) are associated with newborn body composition and later health (e.g. obesity and neurocognitive health).

In the first phase of the study the participants are recruited on postnatal ward after delivery. The umbilical cord blood sample will be collected of all the neonates. After a consent the participants fill in the digital background, food frequency, depression and physical activity questionnaires. If the parents do not give their consent, the umbilical cord blood sample will be destroyed. Body composition of offspring will be assessed within 72 hours after birth. Registry data will be collected.

The second phase of the HeBiCo study is based on the HUS WomensHub treatment path and/or Apotti platform. The second phase of the HeBiCo constitutes of the mother-child pairs (and fathers/spouses) whose pregnancy can be followed from the early pregnancy to the end of the pregnancy through treatment path. Body composition of offspring born in Helsinki Women's Hospital will be assessed within 72 hours after birth.

The future studies will include 1) the intervention studies with digital service concept through WomensHub platform, and 2) the follow-up studies of offspring and parents in later life (to establish e.g. growth trajectories and later metabolic health of offspring).

The first phase of the HeBiCo study was registered 3/2018.

The second phase will be registered now.

ELIGIBILITY:
Inclusion Criteria:

Mothers, fathers/spouses and offspring in Helsinki and Uusimaa Hospital District.

Exclusion Criteria:

Inability to communicate in Finnish language

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The first phase of the Helsinki Birth Cohort (HeBiCo) will be constituted of all the neonates whose body composition at birth can be obtained at Helsinki Women's Hospital, and whose mothers and fathers/spouses fill out the questionnaires after delivery (background, food frequency (FFQ), and depression questionnaires (EPDS, CES-D)).
  In the second phase of HeBiCo, participants will be recruited any time during pregnancy and also at postnatal ward after delivery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neonatal body fat % | Within 72 hours of birth
  Measured with PEA POD Cosmed® Infant Body Composition Assessment system

SECONDARY OUTCOMES:
Newborn weight | Within 2 hours of birth
  Birth weight in kilograms
Newborn height | Within 2 hours of birth
  Birth height in meters
ASQ-3 | 3 months, 1 year and 2 years of age
  Ages and Stages Questionnaire-3
ITSEA | 3 months, 1 year and 2 years of age
  Infant Toddler Social Emotional Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Saila SB Koivusalo, Principal Investigator — Helsinki University Hospital, Women's Hospital
Locations (1):
- HUS Women's hospital, Helsinki Unversity Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No